CLINICAL TRIAL: NCT02184403
Title: Quality of Life After Laser Cordectomy in Early Glottic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Fang Tuan-Jen, Director, Laryngology, Chang Gung Memorial Hospital
Other Study IDs: 99-0579B
Record Dates: First submitted 2014-06-13; First posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Carcinoma of Glottis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Laryngeal cancer is common in the Taiwanese populations. Before early 80's, open laryngectomy was the suggested treatment modality for laryngeal cancer. Patients of laryngectomy lost speech and should communicate by using prosthesis. So after 90's, medical organ preservation by chemoradiation therapy took the place of operation.

Unfortunately, from the recent review, five-year survival rate was decreasing and is even lower than that reported 10 years ago. In 1983-1985 it was 68.1% but decreased to 64.7% in 1992-1999. It is the only cancer type of decreasing survival in 24 index cancers.

Laser resection of laryngeal tumor was first reported by Jako and Strong and widely used in the Europe. Dr Steiner and his colleagues developed a non-en block resection technique made microscopic resection more easily and would not be limited by tumor location or size so much. The investigators used transoral microscopic laser (TLM) in early glottic cancer and reported five-year overall survival as 97%. TLM five-year disease control rate was reported as 85%. There are some reports about TLM in advanced stage laryngeal cancer and overall 5-year survival rate can be achieved as high as 55%. Present project is planning to develop a comprehensive organ preservation protocol based on microinvasive TLM as primary treatment modality for early glottic cancer without neck or distant metastasis. The objects of the project are as followed.

1. Long term outcomes by performing the treatment protocol. The outcome measurements include local control rate, overall and disease specific survival, larynx preservation rate.
2. The difference between surgical samples and pretreatment imaging examination.
3. The role of adjuvant therapy.
4. Management and follow-up in neck metastasis.
5. Searching for risk factors and predictor factors.
6. Adequate salvage treatments in local or regional recurrence.
7. Realizing failure patterns and appropriate follow-up protocol according to it.

DETAILED DESCRIPTION:
Laryngeal cancer is associated with a cure rate from 30 to 90% by primary treatment with irradiation therapy, open surgical excision or microinvasive endolaryngeal surgical excision based on the stages. Prior to advances in endoscopic surgical techniques, radiation therapy with or without chemotherapy offered treatment with less morbidity than open surgical resection. Therefore, throughout the later part of the 20th century, radiation therapy became the standard management for laryngeal cancer.

In the America, the Surveillance, Epidemiology, and End Results (SEER) Program and the National Cancer Data Base (NCDB) data have shown the survival rate of laryngeal cancer decreased in the 1990's. Five-year relative survival for laryngeal squamous cell carcinoma recorded in the NCDB ranged from a high of 68.1% in 1985 to a low of 62.8% in 1993.

Treatment patterns have changed with an increase in nonsurgical management with irradiation alone and with chemoradiation. Radiation or chemoradiation therapies provided a treatment choice to preserve the larynx. However, the increase in nonsurgical management parallels the increase in mortality across the years of study for which survival analysis was performed (1985-1996).

In the past two decades, the evolution of microinvasive TLM surgery makes it possible to eradicate tumors with preserving laryngeal functions. It has been demonstrated that cure rates can be obtained that are comparable with other treatment modalities. In addition, morbidity from treatment by TLM is substantially less than morbidity associated with open surgical techniques and may be the same or less than morbidity associated with radiation or chemoradiation therapy. Therefore, TLM as an initial treatment modality for laryngeal cancer is more commonly practiced.

TLM offers advantages over other forms of treatment. First it can usually be accomplished in a single intervention in early stage of disease- thus decreasing the overall treatment time and cost when compared to radiation therapy. Second, as opposed to open surgical techniques, resection by endoscopic methods does not require a tracheotomy for airway maintenance. Third, rehabilitation time to independent swallowing has been shown in multiple series to be reduced compared with open surgical techniques. And forth, it leaves all opportunities in adjuvant or salvage therapy. Due to these advances, TLM surgery of laryngeal cancer is becoming more widely used in recent years for a focal small lesion and has also been demonstrated to have a comparable survival rate and local control rate in advanced stage to other forms of treatment.

The primary object of the study is to improve the tumor control rate with an organ preservation protocol based on microinvasive TLM surgery. This prospective phase II study is expected to provide evidence in future treatment plan for laryngeal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Early glottic cancer without neck or distant metastasis 2. Cell type : squamous cell carcinoma

Exclusion Criteria:

1. Had previous head and neck radiation or surgery history. 2. Tumor extended beyond subglottis.

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early glottic cancer without neck or distant metastasis and were managed by Laser cordectomy in a tertian referral hospital in Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-05; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Local tumor recurrences | within12 months

SECONDARY OUTCOMES:
Chang from baseline cancer-related quality of life within 12 months. Questionnaire : European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire score C30 | pre-op, post op 1, 3, 6, 12 months
Change of voice quality from baseline. Measured by voice laboratory test including Maximal Phonation Time,S/Z ratio,Fundamental Frequency,Jitter, Shimmer,Harmonics to Noise ratio | pre op, post op 1, 3, 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tuan-Jen Fang, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Linkou District, Taiwan